CLINICAL TRIAL: NCT03890341
Title: A Study in Healthy Female Participants to Investigate the Effect of JNJ-64530440 on the Single-dose of Ethinylestradiol and Drospirenone (Oral Contraceptive), and Midazolam, and the Effect of a High-fat Meal on the Single-dose of JNJ-64530440
Brief Title: Study in Women on the Effect of JNJ-64530440 on Oral Contraceptive and Midazolam, and the Effect of a High-fat Meal on JNJ-64530440
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped due to a strategic decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JNJ-0440-1302; JNJ-0440-1302 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — drospirenone; Ethinyl Estradiol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drospirenone/Ethinylestradiol + Midazolam + JNJ-64530440 (Experimental): Participants will receive single oral dose of drospirenone/ethinylestradiol 3 milligram (mg)/0.02 mg (oral contraceptive [OC]) and midazolam 2 mg with under fed conditions (high fat meal) on Day 1 followed by JNJ-64530440 2,000 mg on Days 6 under fasted conditions ; JNJ-64530440 2,000 mg plus single oral dose of OC and midazolam 2 mg under fed conditions on Day 13; JNJ-64530440 2,000 mg once daily under fed conditions (standard meal) from Days 14 to 18; single oral dose of JNJ-64530440 2,000 mg plus single oral dose of OC and midazolam 2 mg on Day 19 under fed conditions (high fat meal); and JNJ-64530440 2,000 mg once daily under fed conditions (standard meal) on Days 20 to 22.
  Interventions: Drug: Drospirenone/Ethinylestradiol; Drug: Midazolam; Drug: JNJ-64530440

INTERVENTIONS:
Drug: Drospirenone/Ethinylestradiol — A single oral dose of drospirenone/ethinylestradiol 3 mg/0.02 mg (OC) tablets will be administered on Days 1, 13 and 19.
  Other Names: Betadex clathrate
Drug: Midazolam — Midazolam 2 mg will be administered orally on Days 1, 13 and 19.
Drug: JNJ-64530440 — A single oral dose of JNJ-64530440 2,000 mg will be administered on Day 6 and once daily on Days 13 to 22.

SUMMARY:
The purpose of this study is to evaluate the effect of JNJ-64530440 single- and multiple-dose administration on the single-dose pharmacokinetics of drospirenone and ethinylestradiol (oral contraceptive) in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index between 18.0 and 30.0 kilogram per meter square (kg/m^2), extremes included, and a body weight not less than 50.0 kilogram (kg)
* Healthy on the basis of physical examination, medical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the Investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the Investigator
* Must have a negative highly sensitive urine pregnancy test at Day -1 (all participants)
* Must have a negative highly sensitive serum beta-human chorionic gonadotropin pregnancy test at screening (all participants except for postmenopausal participants)
* Must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 90 days after the last study drug administration

Exclusion Criteria:

* Any evidence of heart block or bundle branch block
* History of liver or renal dysfunction (estimated creatinine clearance less than [<] 90 milliliter per minute (mL/min) at screening, calculated by the Modification of Diet in Renal Disease (MDRD) formula), significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Past history of clinically significant cardiac arrhythmias (example [eg], premature ventricular contractions, premature atrial contractions, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* Current human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* Current hepatitis A virus infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or Hepatitis B Virus (HBV) infection (confirmed by Hepatitis B surface antigen [HBsAg]), or Hepatitis C Virus (HCV) infection (confirmed by HCV antibody), or hepatitis E virus infection (confirmed by hepatitis E antibody IgM) at screening

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Drospirenone | Days 1, 13, and 19: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 hours postdose
  Cmax is defined as maximum observed plasma analyte concentration.
Area Under the Plasma Analyte Concentration-Time Curve from Time Zero to Last Quantifiable Concentration Time (AUC [0-Last]) of Drospirenone | Days 1, 13, and 19: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 hours postdose
  AUC(0-Last) is area under the plasma analyte concentration-time curve from time zero to time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinite Time (AUC [0-infinity]) of Drospirenone | Days 1, 13, and 19: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 hours postdose
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); where C(last) is the last observed measurable (non-below quantification limit) concentration.
Maximum Observed Plasma Analyte Concentration (Cmax) of Ethinylestradiol | Days 1, 13, and 19: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 hours postdose
  Cmax is defined as maximum observed plasma analyte concentration.
Area Under the Plasma Analyte Concentration-Time Curve from Time Zero to Last Quantifiable Concentration Time (AUC [0-Last]) of Ethinylestradiol | Days 1, 13, and 19: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 hours postdose
  AUC(0-Last) is area under the plasma analyte concentration-time curve from time zero to time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinite Time (AUC [0-infinity]) of Ethinylestradiol | Days 1, 13, and 19: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 hours postdose
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); where C(last) is the last observed measurable (non-below quantification limit) concentration.

SECONDARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Midazolam | Days 1, 13, and 19: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Cmax is the maximum observed plasma analyte concentration.
Area Under the Plasma Analyte Concentration-Time Curve from Time Zero to Last Quantifiable Concentration Time (AUC [0-Last]) of Midazolam | Days 1, 13, and 19: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  AUC(0-Last) is area under the plasma analyte concentration-time curve from time zero to time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinite Time (AUC [0-infinity]) of Midazolam | Days 1, 13, and 19: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  AUC(0-Last) is area under the plasma concentration-time curve from time zero to time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Cmax of JNJ-64530440 Under Fed Conditions (High-Fat Meal) | Days 13 and 19: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18 and 24 hours)
  Cmax is defined as the maximum observed plasma concentration. Cmax will be assessed under fed conditions (high-fat meal).
Maximum Observed Plasma Concentration (Cmax) of JNJ-64530440 | Days 13 and19: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18 and 24 hours
  The Cmax is the maximum observed plasma analyte concentration.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately up to 70 days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency